CLINICAL TRIAL: NCT03689868
Title: Addressing Parental and Pediatric Anxiety Through Virtual Reality (VR) Intervention in (Limited-English Proficiency) LEP Populations
Brief Title: Limited-English Proficiency (LEP) Virtual Reality (VR) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Samuel Rodriguez, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 46551
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Anxiety; Parents; Language
Keywords: virtual reality
MeSH Terms: conditions — Anxiety Disorders; Language

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental)
  Interventions: Behavioral: Virtual Reality
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Virtual Reality — Virtual Reality headset with calming scenery
  Arms: Virtual Reality

SUMMARY:
The purpose of this study is to determine if non-invasive distracting devices (Virtual Reality headset) are more effective than the standard of care (i.e., no technology based distraction) for preventing anxiety in parental and pediatric populations with limited English proficiency (LEP).

ELIGIBILITY:
Inclusion Criteria:

* Ages 0-99 (Child participants will be ages 0 to 17. Parents of children of any age may also be enrolled)
* Able to consent
* Self-identified as having a limited English proficiency or English-proficiency

Exclusion Criteria:

* People who do not consent
* Significant Cognitive Impairment
* History of Severe Motion Sickness
* Current Nausea
* Seizures
* Visual Problems
* Patients whose children are clinically unstable or require urgent/emergent intervention

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Procedural-Related Anxiety | Duration of intervention, approximately 20-30 minutes
  Validated questionnaires regarding anxiety will be administers pre- and post-intervention (i.e virtual reality) and compared to those in the control arm (i.e no virtual reality)

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] West AM, Bittner EA, Ortiz VE. The effects of preoperative, video-assisted anesthesia education in Spanish on Spanish-speaking patients' anxiety, knowledge, and satisfaction: a pilot study. J Clin Anesth. 2014 Jun;26(4):325-9. doi: 10.1016/j.jclinane.2013.12.008. Epub 2014 Jun 2. PMID 24882604
- [Background] Fabiyi C, Rankin K, Norr K, Shapiro N, White-Traut R. Anxiety among Black and Latina Mothers of Premature Infants at Social-Environmental Risk. Newborn Infant Nurs Rev. 2012 Sep 1;12(3):132-140. doi: 10.1053/j.nainr.2012.06.004. PMID 22962543